CLINICAL TRIAL: NCT00508352
Title: Post-operative Locoregional Irradiation Using Helical Tomotherapy IMRT in the Management of Stage IIb-III Breast Cancer: a Feasibility Study
Brief Title: Post-operative Radiation With IMRT in the Management of Stage IIB-III Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006277-01H
Record Dates: First submitted 2007-07-25; First posted 2007-07-27 (Estimated); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: breast; cancer; locoregional; IMRT; tomotherapy
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Helical tomotherapy (Experimental): Helical tomotherapy IMRT 50 Gy in 25 fractions, daily treatment
  Interventions: Procedure: Helical tomotherapy IMRT

INTERVENTIONS:
Procedure: Helical tomotherapy IMRT — Helical tomotherapy IMRT 50 Gy in 25 fractions, daily treatment

SUMMARY:
Research has shown that treatment with conventional radiation techniques and chemotherapy following mastectomy or breast conserving surgery has resulted in better rates of locoregional control and overall survival in stage IIB-III breast cancer. The current feasibility trial using the most recent advance in radiation therapy, namely helical tomotherapy intensity modulated radiation therapy (HT-IMRT), hopes to improve on the results of conventional radiation by decreasing the amount of radiation-induced toxicity in patients with stage IIb-III breast cancer.

DETAILED DESCRIPTION:
The role of locoregional radiation therapy in the management of stage IIB and III breast cancer has evolved and continues to evolve. The exact role of locoregional radiation, including axillary, supraclavicular and internal mammary nodes is, however, not clear. Radiation-induced toxicity remains a limiting factor to expanding the indications for radiation therapy to axillary and internal mammary nodes in the treatment of stage IIB and III breast cancer. Excellent target coverage and normal tissue sparing of IMRT has been previously demonstrated dosimetrically and clinically. In this feasibility study, patients will receive 50 Gy of radiation therapy in 25 fractions to the chest wall and supraclavicular, axillary and IM nodal areas using HT-IMRT following breast conserving surgery or mastectomy and chemotherapy. Patients will also be eligible for a radiation boost to 12 Gy by HT-IMRT or HDR brachytherapy. It is expected that treatment with HT-IMRT will result in appreciably fewer side-effects following locoregional irradiation due to a reduction in normal tissue irradiation, as compared to conventional radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Surgery with either mastectomy or breast conserving surgery
2. Presence and association of any of the following high risk pathological features present at time of surgery: stage pT3-4 and pN0 and central/medial location of tumour or any pT and pN2 (stage IIB-stage III)
3. All patients will have been treated previously with chemotherapy prior to radiation therapy
4. ECOG performance status of 2 or less

Exclusion Criteria:

1. Prior chest wall/breast or nodal radiation for other malignancies (i.e. Hodgkin disease)
2. HER2+ positive patients
3. Patients with diagnosis of metastatic disease
4. Prior or active malignancy except non-melanoma skin carcinoma within 5 years of the diagnosis of breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Caudrelier, md, Principal Investigator — OHRI
Locations (1):
- The Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Caudrelier JM, Meng J, Esche B, Grimard L, Ruddy T, Amjadi K. IMRT sparing of normal tissues in locoregional treatment of breast cancer. Radiat Oncol. 2014 Jul 22;9:161. doi: 10.1186/1748-717X-9-161. PMID 25052720

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Helical Tomotherapy
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Helical Tomotherapy
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: Years] | 52 [33 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 30

OUTCOME MEASURES:

1. Primary Outcome: Acute Radiation Effects (Less Than 90 Days Post Treatment)
Description: Grade 3 or higher radiation effects(less than 90 days post treatment)
Time Frame: less than 90 days post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Helical Tomotherapy
Number analyzed (Participants) | 30
Participants | 0

2. Primary Outcome: Moderate-late Pulmonary and Cardiac Radiation Effects
Description: Grade 3 or higher moderate-late pulmonary and cardiac radiation effects up to 1 year post radiation
Time Frame: up to 1 year post radiation
Measure: Count of Participants; unit: Participants
Arm/Group | Helical Tomotherapy
Number analyzed (Participants) | 30
Participants | 0

3. Secondary Outcome: Rate of Local Recurrence
Description: Evaluate rate of local recurrence at 5 years
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Helical Tomotherapy
Number analyzed (Participants) | 30
Participants | 0

4. Secondary Outcome: Rate of Regional Recurrence
Description: Evaluate rate of regional recurrence at 5 years
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Helical Tomotherapy
Number analyzed (Participants) | 30
Participants | 0

ADVERSE EVENTS:
Arm/Group | Helical Tomotherapy
All-Cause Mortality (participants affected / at risk) | 6/30
Serious Adverse Events (participants affected / at risk) | 5/30
Other Adverse Events (participants affected / at risk) | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Helical Tomotherapy (N=30)
Distant Recurrent Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No